CLINICAL TRIAL: NCT06945445
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose and Multiple Dose Study of SLN12140 Administered Subcutaneously or Intravenously in Healthy Adult Volunteers
Brief Title: Study of SLN12140 in Healthy Adult Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Linno Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LIN2102-CN101
Record Dates: First submitted 2025-04-10; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SLN12140 (Experimental): a single dose of SLN12140 by subcutaneous (sc) injection:50mg ; a single dose of SLN12140 by subcutaneous (sc) injection:150mg; a single dose of SLN12140 by subcutaneous (sc) injection:450mg ; a single dose of SLN12140 by intravenous(IV) injection:450mg ; a single dose of SLN12140 by subcutaneous (sc) injection:900mg ; a single dose of SLN12140 by subcutaneous (sc) injection:1500mg~1800mg
  Interventions: Drug: SLN12140
- Placebo (Placebo Comparator): Placebo (SLN12140 formulation buffer) will be provided as an injectable solution without active ingredient.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SLN12140 — SLN12140 for sc injection or IV infusion
  Arms: SLN12140
Other: Placebo — Placebo for sc injection or IV infusion
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled phase I clinical study evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of SLN12140 in healthy participants with single subcutaneous/intravenous dose escalation and multiple subcutaneous administrations

DETAILED DESCRIPTION:
This study will include up to 7 different dosing cohorts, with each cohort consisting of 2 groups (SLN12140 group, placebo group). Participants will be randomly assigned in a 3:1 ratio to each of these 2 groups, respectively, within all 7 cohorts, to receive either a single or multiple doses of ALXN1820 SC, a single dose of ALXN1820 IV, or a single or multiple doses of placebo.

The study will be conducted in healthy adult participants .

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in clinical trials and sign written informed consent, and be able to complete the whole trial process according to the requirements of the trial.
2. Persons of any gender, aged between 18 and 65 years old (including the boundary value).
3. Weight: male ≥50kg , female ≥45kg ; Body mass index (BMI) within the range of 19.0 to 28.0 kg/m2 (including cut-off values).
4. Those whose medical history, physical examination, vital signs examination, electrocardiogram examination, laboratory examination indicators, and anteroposterior chest X-ray are all normal or abnormal but non clinically significant as judged by the investigator.
5. Participant has received the following vaccines:

   * Meningococcal polysaccharide vaccine ACYW135 (MPV-ACYW) or meningococcal polysaccharide conjugate vaccine ACYW135 (MPCV-ACYW), given at least two weeks before the first dose and no earlier than within 2 years before the first dose;
   * 13-valent pneumococcal conjugate vaccine (PCV13) or 23-valent pneumococcal polysaccharide vaccine (PPV23) at least two weeks before the first dose, and no earlier than 8 weeks before the first dose of PCV13 and no earlier than 4 years before the first dose of PPV23.
6. Normal or abnormal but no clinical significance with ECG results ,such as QTcF interval ≤450ms (males) and QTcF interval ≤470ms (females); PR interval ≤ 209 ms; The QRS interval ≤ 120 ms.
7. During the study period and within 3 months after the last dose of the study, there is no childcare plan and can take highly effective contraceptive measures and cannot donate sperm or eggs.

Exclusion Criteria:

1. Have cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic or nervous system diseases that affect the absorption, distribution, metabolism or elimination of drugs; or those with disease or medical history that may interfere with the interpretation of study data.
2. Those who have any previous history of Neisseria meningitidis.
3. Those who have a positive skin test for penicillin. Those who have known allergies or contraindications to penicillin or any vaccine ingredients, or who are known to be allergic to the trial drug and any of its ingredients or related preparations, or who have any history of allergies to food, drugs, or allergic diseases or allergies.
4. Those who have or are suspected of having any active viral, bacterial, fungal or parasitic infection, or receiving any anti-infective treatment within 1 month prior to screening.
5. Those with a history of recurrent or chronic infection (such as recurrent upper respiratory tract infection, diarrhea, etc.) within 3 months before screening.
6. Within 1 month prior to screening, have received a live attenuated vaccine, or plan to receive a vaccine during the study (except for vaccinations required for the study).
7. Received drugs that may interact with penicillin V potassium within 7 days or 5 elimination half-lives (whichever is longer) prior to dosing.
8. Those who have any of the following abnormalities in laboratory tests during the screening stage:

   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or alkaline phosphatase (ALP) exceeds the normal range;
   * Total bilirubin (TBIL) ≥ 1.5 times the upper limit of normal (ULN);
   * eGRF (CKD-EPI formula) <90 mL/min/1.73m2;
   * Hemoglobin < lower limit of normal range (LLN).
9. At the time of screening, the results of complement C3 and C4 examinations are lower than the lower limit of the normal reference value range and the abnormalities judged by the investigator to be clinically significant.
10. Immunocompromised, or suffering from at least one of the following underlying diseases:

    * Anatomical or functional asplenia (including sickle cell disease);
    * Congenital complement deficiency (complement factor P deficiency, complement factor B deficiency, or complement factor D deficiency);
    * Acquired complement deficiency;
    * Human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome.
11. Those who are positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, Treponema pallidum antibody (TPPA) and HIV antibody.
12. Those who have donated or lost more than 400 mL of blood or have a history of blood transfusion within 30 days before screening or Day-1.
13. Within 90 days prior to screening or Day-1, the participant has received investigational drug administration, or is currently participating in another clinical study (including the follow-up period).
14. Participants who have used any prescription or over-the-counter medications, any vitamin products, or herbal remedies within 7 days prior to dosing.
15. Those who have any history of intolerance to subcutaneous injection or related injection site scars (surgery, burns, tattoos, etc.) that would affect the evaluation of injectable drug administration.
16. Those who are unwilling or unable to use antibiotic prophylaxis specified in the protocol.
17. A person who falls under any of the following conditions:

    * Professionals at high risk of exposure to meningococcal disease
    * Research, industrial, or clinical laboratory personnel who are at risk of exposure to meningococcals
    * Planned travel to areas where meningococcal is endemic (e.g., India, sub-Saharan Africa, Saudi Arabia) during the study period, or have traveled to these areas within 6 months of the day prior to the start of the study.
18. A current or former drug abuser.
19. Day-1 Positive Drug Abuse Screen.
20. Those who have been an alcoholic within the current period of 3 months or in the past (drinking more than 14 standard units per week. 1 standard unit contains 14 g of alcohol, e.g. 360 mL of beer or 45 mL of spirits with 40% alcohol or 150 mL of wine).
21. Those who have a positive Day-1 alcohol breath test (>0.0mg/100mL).
22. Use of more than 10 cigarettes (or equivalent nicotine-containing products) per week or more than 5 cigarettes (or equivalent nicotine-containing products) per day within 4 weeks prior to screening.
23. Day-1 urine cortinine test positive.
24. Those who have taken a special diet (including dragon fruit, mango, grapefruit, etc.) within 24 hours before administration or have strenuous exercise, or other factors that affect the absorption, distribution, metabolism, and excretion of drugs.
25. Pregnant or lactating female participants or those with a positive pregnancy test.
26. Those who are unable to receive venipuncture, or faint blood and faint needles.
27. Those who are considered by the investigator to have other factors that are not suitable for participating in the trial.

Ages: 18 Days to 65 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SLN12140 | 36 days
  Number of Participants with Adverse Events (AEs) and/or Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics-Cmax | 36 days
  Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics-Tmax | 36 days
  Time at which the maximum plasma concentration (Cmax) occurs
Pharmacokinetics-AUClast | 36 days
  Area under the plasma concentration-time curve from dosing (time zero) to the time of the last measured concentration
Pharmacokinetics-AUCinf | 36 days
  Area Under the Plasma Concentration Versus Time Curve from Zero Extrapolated to Infinity (AUCinf)
Pharmacokinetics-t1/2 | 36 days
  Terminal Elimination Half-Life (t1/2)
Pharmacokinetics-Vd/F | 36 days
  Volume of Distribution (Vd/F)
Pharmacokinetics-CL/F | 36 days
  Total Body Clearance
Pharmacokinetics-λz | 36 days
  Elimination rate constant (λz)
Pharmacokinetics-MRT | 36 days
  Mean retention time (MRT)
Pharmacokinetics-AUC 0-t, sc/AUC 0-t,iv；AUC 0-inf, sc/ AUC 0-inf,iv | 36 days
  Subcutaneous bioavailability-(AUC 0-t, sc/AUC 0-t,iv；AUC 0-inf, sc/ AUC 0-inf,iv)
Pharmacodynamics-CFP | 36 days
  Change From Baseline in Total and Free Complement factor P (CFP)
Pharmacodynamics-AP activity | 36 days
  Change From Baseline in alternative pathway activity (AP)
Pharmacodynamics-CP, LP Activity | 36 days
  Change From Baseline in Classical pathway and Lectin Pathway (CP, LP)
Immunogenicity-ADA, Nab | 36 days
  Anti-drug antibody positive rate (ADA); ADA titer and Neutralizing antibody rate (Nab)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, Doctor of Pharmacy, Principal Investigator — Huashan Hospital; Xiaojie Wu, Doctor of Pharmacy, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - Huashan Hospital, Shanghai, Shanghai Municipality
  - Phase I center of Fudan University Huashan Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No